CLINICAL TRIAL: NCT06899100
Title: Gentle Warriors Academy Program Evaluation
Brief Title: Gentle Warriors Academy Healthy Marriage and Responsible Fatherhood Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Fathers Incorporated (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/42
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Fathers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Services (Experimental): Participants receive 26 hours of Next Level Fatherhood curriculum, 2 hours of child maltreatment workshops, 2 hours of anger management workshops, and 2 hours of optional legitimation workshops. Participants also receive ongoing case management and support services.
  Interventions: Behavioral: Primary Services

INTERVENTIONS:
Behavioral: Primary Services — Participants receive 26 hours of Next Level Fatherhood curriculum, 2 hours of child maltreatment workshops, 2 hours of anger management workshops, and 2 hours of optional legitimation workshops. Participants also receive ongoing case management and support services.

SUMMARY:
The purpose of this descriptive study is to explore whether there is an association between participation in the Gentle Warriors Academy and improvements in outcomes related to parenting, co-parenting, and parental well-being. Participants are surveyed at program entry, program exit, and 12 months following program enrollment, and changes in participant attitudes and behaviors are assessed over time.

DETAILED DESCRIPTION:
This study is a descriptive evaluation of the Gentle Warriors Academy program offered to fathers in the Atlanta metropolitan area. Program participants are informed about the study and asked to provide consent to participate in the evaluation of the program. Consenting participants complete surveys at program enrollment, program exit, and 12 months after program enrollment, and survey data is used to determine if the program is associated with short-term and long-term changes in attitudes and behaviors among participants. Changes in parenting attitudes and parental well-being are assessed by comparing survey answers before and after participating in 26 hours of the Next Level Fatherhood primary curriculum. Changes in behaviors related to parenting and co-parenting are assessed from program entry to 12 months post-enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older)
* Father/father figure
* With children under age 16
* Reside in Metro Atlanta area

Exclusion Criteria:

* Minor (under the age of 18)
* Not a father/father figure
* Children older than 16 years old
* Reside outside of Metro Atlanta area

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 731 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2025-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation and Research
Locations (1):
- Fathers Incorporated, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Services
Started | 731
Completed | 731
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Services
Number analyzed (Participants) | 731
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 730
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 33.87 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 731
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 29
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 7
  Black or African American | 666
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: 1) Healthy Parenting Attitudes Measurement #1
Description: Will participants report significantly healthier parenting attitudes after completing primary workshops, as compared to responses at program enrollment?
  Items measured include:
  Parenting attitudes measured with:
  7 items - frequency of feelings about participant's youngest child (categorical, 5-point scale)
  Measured on the parenting attitudes scale #1 as:
  1 = always, 2 = often, 3 = sometimes, 4 = rarely, 5 = never
  The construct is created by adding all 7 scores together and dividing by 7. The higher the score on a scale of 1-5, the better the outcome. The lower the score, the worse the outcome.
  Maximum score: 5.0, minimum score: 1.0
Time Frame: baseline and program exit at 10 weeks post-enrollment
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 288
score on scale
  mean at baseline | 4.66 (.351)
  mean at program exit at 10 weeks post-enrollment | 4.656 (.346)

2. Primary Outcome: 2) Healthy Parenting Behaviors Measurement #1
Description: Will participants report significantly healthier parenting behavior one year after enrolling in the program, as compared to responses at baseline?
  Items measured include:
  Parenting behavior measured with:
  11 items - frequency of key behaviors with participant's youngest child (categorical, 5-point scale)
  Measured on the parenting behavior scale #1 as:
  1 = never, 2 = 1 to 2 days per month, 3 = 3 or 4 days per month, 4 = 2 or 3 days per week, 5 = every day or almost every day
  The higher the rating, the better the score.
  The construct is created by adding all 11 scores together and dividing by 11. The higher the score on a scale of 1-5, the better the outcome. The lower the score, the worse the outcome.
  maximum score: 5.0, minimum score: 1.0
Time Frame: Time frame: change from baseline in parenting behaviors (interactions with child) from enrollment to 1 year post-enrollment.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 123
score on scale
  mean at baseline | 3.85 (1.03)
  mean at follow-up | 3.94 (0.93)

3. Primary Outcome: 3) Healthy Co-parenting Behaviors Measurement #1
Description: Will participants report significantly healthier co-parenting behavior one year after enrolling in the program, as compared to responses at baseline?
  Items measured include:
  11 items: frequency of agreement with key co-parenting behaviors (categorical, 5-point scale)
  Measured on the co-parenting behavior scale #1 as:
  1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree
  The construct is created by adding all scores together and dividing by 11. The higher the score on a scale of 1-5, the better the outcome. The lower the score, the worse the outcome.
Time Frame: change from baseline in co-parenting behaviors (interactions with co-parent) from enrollment to 1 year post-enrollment.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 442
score on scale
  mean at baseline | 2.90 (1.10)
  mean at follow-up | 2.94 (1.00)

4. Primary Outcome: 4) Parent Wellbeing Measurement #1
Description: Will participants report significantly higher parental wellbeing after completing primary workshops, as compared to responses at program enrollment?
  1 item: frequency of feeling overwhelmed by parenting responsibilities (categorical, 4-point scale)
  1 = never, 2 = hardly ever, 3 = sometimes, 4 = often
  The lower the number, the better the score. Maximum score=4.0, minimum score=1
Time Frame: change from baseline in parental wellbeing (feelings about parenting) from enrollment to program exit (10 weeks).
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 129
score on scale
  mean at baseline | 2.74 (1.06)
  mean at follow-up | 3.02 (0.97)

ADVERSE EVENTS:
Time Frame: 1 year through study completion
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definitions.
Arm/Group | Primary Services
All-Cause Mortality (participants affected / at risk) | 0/731
Serious Adverse Events (participants affected / at risk) | 0/731
Other Adverse Events (participants affected / at risk) | 0/731

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT06899100/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT06899100/SAP_001.pdf